CLINICAL TRIAL: NCT02018341
Title: A Randomized Double-blind Placebo Controlled Homeopathic Pathogenetic Trial (HPT) on Healthy Volunteers Proving XX in the Potency of 30C, "The Homeogenomic Trial"
Brief Title: The Homeogenomic Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, James Taylor, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 44817
Record Dates: First submitted 2013-06-20; First posted 2013-12-23 (Estimated); Last update posted 2013-12-23 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Assessment of biologic activity of a homeopathic remedy
MeSH Terms: interventions — Homeopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- homeopathic remedy in 30C potency (Experimental): 5 lactose globules containing a commonly used homeopathic remedy in the potency of 30C will be administered twice daily for 3 days
  Interventions: Other: homeopathic remedy in 30C potency
- placebo (Placebo Comparator): 5 lactose globules without any homeopathic remedy will be administered twice daily for 3 days
  Interventions: Other: Placebo

INTERVENTIONS:
Other: homeopathic remedy in 30C potency
  Arms: homeopathic remedy in 30C potency
Other: Placebo
  Arms: placebo

SUMMARY:
A randomized double-blind placebo controlled homeopathic pathogenetic trial (HPT) will be carried out on 30 healthy adult volunteers. The remedy used for the proving will be administered in a potency of 30C. The remedy being used is a common homeopathic remedy commercially available in the US, but the exact remedy is not disclosed to participants.The purpose of the proving is twofold: 1) to determine if there is a difference in symptoms between those receiving an active versus placebo medicine, and 2) to see if there is a difference in gene expression between those who receive the homeopathic remedy or placebo. It is hypothesized that participants receiving the active medication will have more symptoms characteristic of the remedy and have specific patterns of gene expression in whole blood that are different from those in placebo recipients. Participants will record symptoms in a diary for 3 days prior to administration of study medications, during 3 day of its administration and for 3 days following completion of the study medication. Blood will be drawn for gene expression studies on the day that the study medication is started and again after taking the study medication for approximately 48 hours. An additional, optional blood draw for possible future analysis of gene expression will be done at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Read and Speak English

Exclusion Criteria:

* Acute illness in last 7 days
* Chronic illness requiring daily medication
* Use of homeopathic remedy within 4 weeks
* Use of homeopathic remedy of 200C potency in past 2 months
* Women who are pregnant or breastfeeding an infant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Characteristic symptoms | 6 days
  Symptoms that occur in participants that are characteristic of the homeopathic remedy being used in the study
gene expression | 2 days
  Changes in whole blood gene expression from just prior to beginning study medication until 48 hours after beginning study medication

SECONDARY OUTCOMES:
gene expression in sensitive provers | 2 days
  gene expression in participants receiving active study medication and who are classified as sensitive provers based on review of their symptoms will be compared to gene expression in placebo recipients.

CONTACTS AND LOCATIONS:
Overall Officials: James A Taylor, MD, Principal Investigator — University of Washington
Locations (1):
- Bastyr University, Kenmore, Washington, United States